CLINICAL TRIAL: NCT02825485
Title: Minimizing the Utilization of Voiding Cystourethrography for Patients With Antenatal Hydronephrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Nora Kern, MD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 19030
Record Dates: First submitted 2016-06-23; First posted 2016-07-07 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Antenatal Hydronephrosis; Post-natal Hydronephrosis

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control Group (Other): The control patients will be the patients with antenatal hydronephrosis who get a routine VCUG to evaluate for vesicoureteral reflux, as part of routine care.
  Interventions: Procedure: Voiding cystourethrogram
- Observation Group (No Intervention): Receives no intervention

INTERVENTIONS:
Procedure: Voiding cystourethrogram
  Arms: Control Group

SUMMARY:
It has previously been found that there is no correlation between degree of hydronephrosis and presence of reflux; however this is oftentimes the criteria physicians use to obtain a VCUG.

DETAILED DESCRIPTION:
Investigators conducted a previous retrospective study to evaluate other possible findings on ultrasound that may better predict reflux. Investigators found that if a postnatal ultrasound showed any of the three findings of hydroureter, duplication or dysmorphic kidney, then the odds ratio of detecting reflux was 8.07 (95%CI 3.86, 16.87). The purpose of this study is to perform a randomized prospective study to validate this retrospective study. Investigators hypothesis is that patients with hydronephrosis alone will be more likely to have negative VCUG studies; hence obtaining a VCUG for this indication may not be warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of antenatal hydronephrosis who have a post-natal ultrasound demonstrating hydronephrosis alone and no other abnormalities

Exclusion Criteria:

* Patients with a post-natal ultrasound demonstrating bilateral hydronephrosis
* Patients with a history of posterior urethral valve or when a valve is suspected
* Patients who have hydronephrosis on ultrasound as well as other findings including duplication, hydroureter, dysmorphic kidneys, or bladder abnormalities

Ages: 0 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Development of UTIs | Through study completion, an average of 4 years

SECONDARY OUTCOMES:
The rate of reflux detected on VCUGs | Through study completion, an average of 4 years
Rate of resolution of hydronephrosis | Through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Health System, Pediatric Urology, Battle Bldg, Charlottesville, Virginia, United States